CLINICAL TRIAL: NCT02988063
Title: Effect of Polidocanol Endovenous Microfoam (PEM) Treatment of Superficial Axial and Tributary Vein Reflux on Improvement of Wound Healing in Venous Leg Ulcers (VLUs)
Brief Title: Effect of PEM Treatment of Superficial Axial and Tributary Vein Reflux on Improvement of Wound Healing in VLUs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: OhioHealth (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Raghu Kolluri, Vascular Medicine Physician/System Medical Director, OhioHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OH1-16-00664
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Leg Ulcer; Veins, Varicose; Venous Ulcer; Reflux; Venous Reflux; Venous Leg Ulcer; Varicose Veins; Varicose Ulcer; Varicose Veins Leg
Keywords: Varithena; Polidocanol Endovenous Microfoam
MeSH Terms: conditions — Leg Ulcer; Varicose Veins; Varicose Ulcer; Gastroesophageal Reflux | interventions — Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Compression plus PEM (Experimental): Patients will receive 4-5 weeks of compression therapy, followed by treatment with 1% polidocanol endovenous microfoam (PEM) and 12 additional weeks of compression therapy. If the treating physician determines that the vein is not closed after a subjective assessment of vein patency via standard-of-care limited duplex imaging, patients will be re-treated with PEM on Day 4.
  Interventions: Drug: Polidocanol Endovenous Microfoam (PEM)

INTERVENTIONS:
Drug: Polidocanol Endovenous Microfoam (PEM) — Polidocanol endovenous microfoam (PEM) is a sclerosing agent indicated for the treatment of incompetent great saphenous veins, accessory saphenous veins, and visible varicosities of the great saphenous vein system above and below the knee. PEM improves the symptoms of superficial venous incompetence and the appearance of visible varicosities.
  Other Names: Varithena

SUMMARY:
This study evaluates the addition of polidocanol endovenous microfoam (PEM) to compression therapy to determine effectiveness in improving the healing of venous leg ulcers (VLUs) in adults with severe venous disease of the great saphenous vein (GSV). All participants will receive treatment with Varithena and compression therapy.

The purpose of this study is to assess whether the use of PEM to correct superficial axial and varicose vein reflux is effective in improving healing of VLUs, over treatment with compression alone.

DETAILED DESCRIPTION:
Compression therapy and polidocanol endovenous microfoam (PEM) are both used for the treatment of venous leg ulcers (VLUs), but they do so by different mechanisms.

Compression therapy applied by a wound care professional has been demonstrated to improve healing rates in patients with existing VLUs and to reduce ulcer recurrence, and is used consistently by treating physicians. Compression therapy consists of hosiery, tubular bandages and bandage systems comprising two or more components, which provide graduated compression to the lower limb in order to improve venous return and to reduce edema.

Polidocanol endovenous microfoam (PEM) is an injectable foam medication that is used to treat symptoms of venous disease, including venous leg ulcers (VLUs). The medication ("polidocanol") is in the foam ("endovenous microfoam"). PEM is injected through a catheter or by direct injection into the malfunctioning vein. The foam fills and treats the desired section of the vein, thereby collapsing the diseased vein. When the malfunctioning vein collapses, the microfoam is deactivated and blood flow shifts to healthier veins nearby.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Active VLU with a CEAP classification of C6
* Non-healing VLU ≥ 1 month but not greater than 24 months
* In the case of more than one ulcer, the largest ulcer (compliant with study criteria) will be chosen as the study ulcer and treated in the study. Other ulcerations, if present on the same leg must be at least 2cm apart from the study ulcer.
* Demonstrable GSV insufficiency (as per the Society for Vascular Surgery [SVS] and the American Venous Forum [AVF] Guidelines) via venous insufficiency study (VIS) (11)
* VLU considered non-healing (clinically defined as ≤70% wound improvement) after a 4-5 week run-in period with compression therapy
* Venous leg ulcer size ≥ 2cm2 within the great saphenous distribution and must be visualized in one plane to allow for image collection of the entire wound in one photo by the Silhouette device.
* The ulcer must extend through both the epidermis and dermis, with no exposed tendon or bone
* The ulcer must be located below the knee
* The ulcer bed must have some viable tissues with some granulation tissue
* Able to tolerate effective compression bandaging
* Patients able to walk independently with or without mobility aids
* Ability to comprehend and sign an informed consent document and complete study questionnaires in English
* Able and willing to attend all follow up visits

Exclusion Criteria:

* Age < 18 years old
* Small saphenous vein (SSV) distribution VLUs
* Patients who had previously received interventions for underlying venous disease or prior VLU treatments that would not be considered to be conservative, in the opinion of the principal investigator
* Exposed bone, tendon, or fascia
* Deep vein reflux unless clinically insignificant in comparison to superficial reflux
* Patients with leg ulceration etiology other than venous insufficiency
* Severe rheumatoid arthritis
* History of radiotherapy to the ulcer site
* Uncontrolled congestive heart failure (left or right sided heart failure)
* Receiving corticosteroids or immune suppressive therapy
* Active clinical infection of the ulcer site, however, patients may be entered into the study after successful treatment of infection
* History of collagen vascular disease
* History of known malnutrition (albumin <3.0 g/dL)
* History of known uncontrolled diabetes [hemoglobin A1c (HgbA1c) >8.0%]
* History of known arterial insufficiency [ankle-brachial index (ABI) <0.7, transcutaneous oxygen (tcpO2) <35 mmHg, or toe-brachial index (TBI) <0.4]
* Signs of cellulitis, osteomyelitis, or necrotic or avascular ulcer bed(s)
* Active sickle cell disease
* Patients diagnosed with DVT or phlebitis in the affected limb in the last 6 months, or with acute pulmonary embolism (PE) in the last 6 months (contraindication to PEM)
* Known allergic response to polidocanol or heparin, including history of heparin-induced thrombocytopenia, and/or multiple allergic reactions (contraindication to PEM)
* Chronic renal disease, if deemed by the principal investigator to be severe enough to interfere with wound healing
* Known active or recurrent cancer, or currently receiving chemotherapy or radiation therapy
* Poorly controlled asthma
* Pulmonary edema
* Major surgery, prolonged hospitalization, or pregnancy within 3 months of screening
* Minor surgery within 1 month of screening
* Current alcohol or drug (illicit or prescription) abuse
* Pregnant or lactating women
* History of stroke
* Unable to comply with the procedures described in the protocol
* Unable to comply with compression therapy recommendations
* Unable to give informed consent
* Non-English speaking
* Enrolled in a clinical evaluation for another investigational wound-care device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Ulcer healing rate | 12 weeks
  We will determine the change in ulcer healing rate following PEM treatment. Ulcer healing rate will be measured as the relative weekly change in ulcer perimeter (cm) from baseline, until either until fully healed, or up to the final active study visit at 12 weeks (whichever is sooner). Pre-treatment healing rate will be measured as the relative change in ulcer perimeter (cm) from baseline per week over the 4-5 week run-in period.

SECONDARY OUTCOMES:
Proportion of patients who successfully heal | 12 weeks
  We will determine the proportion of patients who successfully heal by 12 weeks. "Successful" healing will be defined as complete resolution of the ulcer (0 cm), with a lack of disruption of the epithelium at the ulcer site.
Proportion of patients who experience symptomatic pulmonary embolism and deep vein thrombosis (PE and DVT, respectively) and other drug-related adverse events (AEs) | 12 weeks
  We will determine the proportion of patients who experience symptomatic pulmonary embolism and deep vein thrombosis (PE and DVT, respectively) and other drug-related adverse events (AEs) at 12 weeks (or the last active study visit if healed prior to 12 weeks). The most commonly reported drug-related AEs (occurring in ≥3% of patients) include pain/discomfort in extremity, infusion site thrombosis (retained coagulum), injection site hematoma or pain, and superficial thrombophlebitis.

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Kolluri, MD, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth Riverside Methodist Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No